CLINICAL TRIAL: NCT04563754
Title: The Effectiveness of High Resolution Microendoscopy (HRME) in High Grade Intraepithelial Lesions (HSIL) Diagnosis for People Living With HIV
Brief Title: The Effectiveness of High Resolution Microendoscopy for People Living With HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); William Marsh Rice University (Other); University of California, San Francisco (Other); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sharmila Anandasabapathy, Professor of Medicine, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H-44616 Anal HRME
Record Dates: First submitted 2020-03-10; First posted 2020-09-24 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Anal High Grade Squamous Intraepithelial Lesion
MeSH Terms: interventions — Proflavine

STUDY DESIGN:
Intervention Model Description: This is a single-arm study where all subjects will receive both standard of care HRA (High resolution anoscopy) and experimental mHRME imaging.
Masking Description: No masking will be used in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mHRME (Experimental): 5-10 ml of proflavine hemisulfate (0.01%) will be applied on the anal epithelium. The mHRME will then be inserted and imaging of abnormal tissues will be performed.
  This is a single-arm study where all subjects will receive both standard of care HRA (High resolution anoscopy) and experimental mHRME imaging.
  Interventions: Diagnostic Test: mHRME (Mobile High resolution microendoscope); Drug: Proflavine Hemisulfate; Diagnostic Test: High resolution anoscopy

INTERVENTIONS:
Diagnostic Test: mHRME (Mobile High resolution microendoscope) — Standard of care (SOC) high-resolution anoscopy (HRA) with Lugol's iodine will be performed. The unstained (abnormal) area will be evaluated with mHRME for optical biopsy diagnosis:
  1. contrast agent will be applied to anal epithelium (5-10 ml of proflavine hemisulfate (0.01%)),
  2. the mHRME will then be inserted and imaging of abnormal tissues will be performed. This will add 2 to 6 minutes per procedure.
  This is a single-arm study where all subjects will receive both SOC HRA and experimental mHRME imaging.
Drug: Proflavine Hemisulfate — Contrast agent will be applied to anal epithelium (5-10 ml of proflavine hemisulfate (0.01%)) to use with the mHRME
Diagnostic Test: High resolution anoscopy — Standard of care (SOC) HRA with Lugol's iodine will be performed.

SUMMARY:
The investigators have developed a portable, battery-operated, mobile high-resolution microendoscope (mHRME) that provides subcellular images of the anal epithelium, delineating the cellular and morphologic changes associated with neoplasia. The investigators' central hypothesis is that this 'optical' approach will increase the efficiency, clinical impact, and cost-effectiveness of the current standard of high-resolution anoscopy(HRA)-guided biopsy, thus facilitating usage by less-experienced clinicians in community-based or low-resource settings. To validate this, the investigators will conduct a study to determine the efficiency and diagnostic characteristics of the mHRME 'optical biopsy' approach versus the current standard of HRA-based tissue biopsy. Successful results will allow for improved efficacy and resource utilization for cancer screening in people living with HIV for anal cancer and other epithelial cancers including the cervix, oral cavity, bladder, and GI tract.

DETAILED DESCRIPTION:
The investigators' central hypothesis is that using mHRME plus three-dimensional (3D) mapping as a diagnostic tool will improve the accuracy and efficiency of HSIL diagnoses. Additionally, the investigators hypothesize that the sensitivity (SN) specificity (SP), positive predictive value (PPV), and negative predictive value (NPV), as well as the receiver operating characteristic (ROC) curve for the identification of neoplasia on a per biopsy and per patient basis will be high. The investigators will first compare the HRA-directed biopsy (as the gold standard) to the results of the mHRME HSIL diagnosis. The SN of mHRME diagnosis in the detection of HSIL will be estimated with the binomial proportion of study participants who are positive for HSIL on HRA-guided biopsy at two thresholds of histology thresholds which are: 1) Anal intraepithelial neoplasia (AIN) 2+ threshold, and 2) AIN3+ threshold. SP will be estimated as the proportion of study participants who are negative for HSIL on HRA-guided biopsy at both thresholds. PPV and NPV will be estimated using the binomial proportion and 95% confidence interval (CI). In addition, Cohen's kappa statistic and ROC curves will be generated if patient characteristics such as low Clusters of differentiation 4 (CD4) count, combined antiretroviral treatment (cART) utilization, or high HIV viral load impact the determination of SN and SP. SN and SP of mHRME-based HSIL diagnosis will be estimated on a per lesion and per patient basis with 95% CI and compared by McNemar's test. A generalized linear model for logistic regression with multiple correlated outcomes will compare SN and SP of each method on a per biopsy and per patient basis.

Primary Objective:

To determine if the mHRME plus 3D mapping improves the accuracy of anal HSIL diagnosis compared to the gold standard of histologic diagnosis of HSIL by HRA-guided biopsy.

Secondary Objectives:

Determination whether HRME changes the decision to perform biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Consentable patients with documented HIV disease
* Either: 1) previously documented HSIL or 2) abnormal anal cytology within the past 2 years
* Ages 18 years and older
* Seen at the Baylor-affiliated Thomas Street Clinic (TSC), Mount Sinai Hospital and affiliated clinics

Exclusion Criteria:

* Unable to undergo routine anoscopy
* Allergy or prior reaction to the fluorescent contrast agent Proflavine or Iodine
* Unable to give informed consent
* Current or prior history of Invasive Anal Cancer
* Known permanent or irreversible bleeding disorder, or other hematologic disorder that in the opinion of the investigator would place the patient at increased risk for adverse outcome from the procedure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmilla Anandasabapathy, MD, Principal Investigator — Baylor College of Medicine; Elizabeth Y Chiao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Brenes D, Kortum A, Carns J, Mutetwa T, Schwarz R, Liu Y, Sigel K, Richards-Kortum R, Anandasabapathy S, Gaisa M, Chiao E. Automated In Vivo High-Resolution Imaging to Detect Human Papillomavirus-Associated Anal Precancer in Persons Living With HIV. Clin Transl Gastroenterol. 2023 Feb 1;14(2):e00558. doi: 10.14309/ctg.0000000000000558. PMID 36729506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two anal dysplasia clinics: Tisch Cancer Institute Mount Sinai in New York, NY, and Thomas Street Health Center in Houston, TX. At Tisch Cancer Institute Mount Sinai, participants were recruited between July 30, 2019, and September 28, 2021. At Thomas Street Health Center, participants were recruited between December 8, 2021, and March 28, 2023. Participants were consented and screened for eligibility at time of presentation to the two recruitment sites.
Groups:
- Tisch Cancer Institute Mount Sinai: Participants enrolled in the Tisch Cancer Institute Mount Sinai.
- Thomas Street Health Center: Participants enrolled in the Thomas Street Health Center, excluding the first 18 participants used as test subjects.
- Training Set Cohort: The first 18 participants enrolled in the Thomas Street Health Center as test subjects.
Period: HRME Procedure
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
Started | 79 | 66 | 18
Completed | 68 | 60 | 0
Not Completed | 11 | 6 | 18
Not completed — No HRA and/or HRME data due to technical difficulties or quality control issues with HRME imaging | 11 | 6 | 0
Not completed — Optimization/validation of 3D imaging and HRME | 0 | 0 | 18
Period: Follow up
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
Started | 79 | 66 | 18
Completed | 18 | 13 | 13
Not Completed | 61 | 53 | 5
Not completed — Lost to Follow-up | 61 | 23 | 5
Not completed — Death | 0 | 2 | 0
Not completed — Ongoing | 0 | 28 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort | Total
Number analyzed (Participants) | 79 | 66 | 18 | 163
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45.0 [36.0 to 56.0] | 48.0 [36.0 to 57.0] | 50.5 [37.0 to 59.0] | 47.0 [36.0 to 56.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 2 | 11
  Male | 75 | 61 | 16 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 36 | 12 | 82
  Not Hispanic or Latino | 45 | 30 | 6 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 8 | 0 | 0 | 8
  Black or African American | 24 | 26 | 4 | 54
  White | 33 | 12 | 6 | 51
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 25 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Performance Characteristics: Sensitivity (SN), Specificity (SP), Positive Predictive Value (PPV) and Negative Predictive Values (NPV)
Description: The primary outcome of this study is to measure the operating characteristics including SN, SP, PPV and NPV comparing the physician- and algorithm- guided HRME-based image compared to the Lugol's- guided physician diagnosis of HSIL during HRA. Gold standard consensus pathology was used and pathology data needs to be obtained, verified, and entered.
Time Frame: 1 day
Population: The training set cohort (n=18) was used to optimize and develop the automated algorithms assessed for primary and secondary outcomes in the actual clinical study. In both the training set cohort and the clinical study, subjects unable to complete the HRME examination or undergo evaluation with the automated algorithm (n=26) were excluded. The remaining 137 evaluable subjects had images assessed by the algorithm and were analyzed separately by study site and the training set cohort.
Measure: Number (95% Confidence Interval); unit: percentage of biopsies
Units Other Than Participants: Biopsies
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
Number analyzed (Participants) | 68 | 60 | 9
Number analyzed (Biopsies) | 101 | 126 | 20
percentage of biopsies
  HRA - SN | 90.0 [76.3 to 97.2] | 76.9 [56.4 to 91.0] | 100.0 [66.4 to 100.0]
  HRA - SP | 65.6 [52.3 to 77.3] | 48.0 [37.9 to 58.2] | 90.9 [58.7 to 99.8]
  HRA - PPV | 63.2 [49.3 to 75.6] | 27.8 [17.9 to 39.6] | 90.0 [55.5 to 99.7]
  HRA - NPV | 90.9 [78.3 to 97.5] | 88.9 [77.4 to 95.8] | 100.0 [69.2 to 100.0]
  HRME - SN | 90.0 [76.3 to 97.2] | 92.3 [74.9 to 99.1] | 100.0 [66.4 to 100.0]
  HRME - SP | 67.2 [54.0 to 78.7] | 68.0 [57.9 to 77.0] | 100.0 [71.5 to 100.0]
  HRME - PPV | 64.3 [50.4 to 76.6] | 42.9 [29.7 to 56.8] | 100.0 [66.4 to 100.0]
  HRME - NPV | 91.1 [78.8 to 97.5] | 97.1 [90.1 to 99.7] | 100.0 [71.5 to 100.0]

2. Secondary Outcome: Procedure Efficiency
Description: Diagnostic yield: The number of neoplastic biopsies/total number of biopsies obtained in patients who received biopsies.
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of biopsies
Units Other Than Participants: Biopsies
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
Number analyzed (Participants) | 68 | 60 | 9
Number analyzed (Biopsies) | 101 | 126 | 20
percentage of biopsies | 39.6 [30.0 to 49.8] | 20.6 [13.9 to 28.8] | 45.0 [23.1 to 68.5]

3. Secondary Outcome: Procedure Time
Description: Total procedure time (HRA+HRME+biopsies) vs HRME time alone
Time Frame: 1 day
Population: The training set cohort (n=18) was used to optimize and develop the automated algorithms assessed for primary and secondary outcomes in the actual clinical study. In both the training set cohort and the clinical study, subjects who did not have both the procedure start and end times recorded were excluded (n=10). The remaining 153 subjects were analyzed separately by study site and the training set cohort.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
Number analyzed (Participants) | 77 | 61 | 15
minutes
  Total procedure time | 8 [6 to 13] | 12 [10 to 15] | 17 [13 to 18]
  HRME time | 2 [1 to 3] | 4 [3 to 5] | 5 [4 to 6]

ADVERSE EVENTS:
Time Frame: Subjects will be contacted for adverse events 2 and 30 days from procedure. Patients with abnormal clinical findings will be followed until the condition resolves or stabilizes. Adverse events or serious adverse events that occur during the follow-up period will be recorded regardless of relatedness to the study procedure.
Description: We will use Common Terminology Criteria for AE v5.0. Serious adverse events will count as Grade 3 (Severe or Medically Significant, but not Immediately Life Threatening: Hospitalization or Prolongation of Hospitalization Indicated; Disabling; Limiting Self Care ADL), Grade 4 (Life-threatening consequences; urgent intervention indicated) or Grade 5 (Death related to AE).
Arm/Group | Tisch Cancer Institute Mount Sinai | Thomas Street Health Center | Training Set Cohort
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/66 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/66 | 0/18
Other Adverse Events (participants affected / at risk) | 0/79 | 0/66 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04563754/Prot_SAP_004.pdf
  • Informed Consent Form (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04563754/ICF_003.pdf